CLINICAL TRIAL: NCT02572037
Title: Research and Clinical Value of New Classification for Premature Ejaculation:Multi-Center Research
Brief Title: Research and Clinical Value of New Classification for Premature Ejaculation: Multi-Center Research
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Baibing Yang, Resident of Nanjing Drum Tower Hospital, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: BL2014001
Record Dates: First submitted 2015-09-27; First posted 2015-10-08 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation; Dapoxetine; local anaesthetics; nerve electrophysiology
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: Penile sensory hyperexcitability: Latencies of GPSEP and/or DNSEP of them are abnormal. They will receive treatment of Compound Lidocaine Cream-a kind of local anaesthetics that is widely used to treat PE.
- Group II: Sympathetic hyperexcitability: Latency of PSSR are abnormal.They will be treated with Dapoxetine(Priligy)-a kind of selective serotonin reuptake inhibitor(SSRI) which has been shown effective to PE.
- Group III: Mixed type: Both Latencies of GPSEP and/or DNSEP and Latency of PSSR are abnormal.They will receive both Compound Lidocaine Cream and Dapoxetine.
- Group IV: Others: Both Latencies of GPSEP, DNSEP and Latency of PSSR are normal.They will receive further tests. (This group is not the main objects to be observed in this study.)

SUMMARY:
An observational study on the effect of new classification for premature ejaculation.

DETAILED DESCRIPTION:
Premature ejaculation (PE) is one of the the most common male sexual dysfunctions and it has negative impacts on people's quality of life. According to the time that PE syndromes come out, PE is clinically divided to primary PE , which appear from the first sex ,and secondary PE ,which occurred after a period of normal ejaculation. This method of classification make little sense for treatment. In 2008, PE was divided into four types: primary PE, secondary PE, natural variable PE and premature-like ejaculatory dysfunction , and different types of premature ejaculation have their corresponding treatment. Both method of classification are based on the subjective feelings of patients, then whether certain objective test can be used to help diagnosing premature ejaculation? The drug treatment of PE mainly includes local anesthetics and selective 5- serotonin reuptake inhibitor (SSRI), and the selective penile dorsal nerve block is the most used surgery. But the efficacy of dapoxetine(a new SSRI for PE) and local anesthetics is only about 60-70% and 60%, respectively, while the efficacy of surgery is not exact without a standard surgical indication. We suppose that there may be different subtypes of the nerve of patients with premature ejaculation may exist in, which corresponds to a specific treatment.

In previous study, the investigators studied the somatic sensory pathway and autonomic nerve function of patients with premature ejaculation, and found that they were characterized by different neural electrophysiological characteristics. About 60% patients with primary PE show hypersensitivity of penis, and the efficacy of local anesthetics or selective penile dorsal nerve block for them reached 90%. While SSRI can reduce the excitability of the sympathetic nervous system in patients with PE, and the effect of this drug on patients with Sympathetic hyperexcitability is better than those without Sympathetic hyperexcitability. Thus doctors here have already been dividing patients who only suffer from PE(no other diseases mentioned in exclusion criteria)into 4 groups according to the results of nerve electrophysiological examination and give corresponding treatment: 1. Penile sensory hyperexcitability Group, using local anaesthetics(compound lidocaine cream)to treat; 2. Sympathetic hyperexcitability Group: using selective serotonin reuptake inhibitor(SSRI)(Dapoxetine) to treat. 3. Mixed type Group: both Penile sensory hyperexcitability and Sympathetic hyperexcitability: Combined use of two treatments above. 4. Other Group: result of nerve electrophysiological examination is normal: this group of patients will receive further examination to figure out the reason. This pattern of treatment has been used in clinical practice for years.

In this research, the investigators will systemically observe the result of this classification and treatment for 12 weeks. Patients will be asked for participating in this research. The questionnaires(IELT,PEDT,PEP) can be filled in when visited or online about every 4 weeks. If he refused , he would still receive the classified treatment but not enrolled in this research. After treatment of 12 weeks, the investigators will measure the change of IELT, PEDT, PEP, nerve electrophysiological examination and CGIC, then compare the efficacy of the treatment to that has been reported before. If anyone do not want to continue the treatment, he could quit from this research. Software SPSS17.0 will be used for data analysis. The age, height, weight, quantity table, the latency and amplitude of each group will be expressed by the mean add or subtract standard deviation. Quantitative data comparison among groups was analyzed by single factor variance analysis (one-way ANOVA and LSD), comparison of rate using x2 test, comparison of before and after treatment compared with paired t test. P<0.05 showed statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 18 and 60;
2. Men in stable heterosexual, monogamous relationships >6 months;
3. Symptom of PE: Ejaculation that always or nearly always occurs prior to or within 2 minute of vaginal penetration from the first sexual experience; the inability to delay ejaculation; and negative personal consequences, such as distress, bother, frustration, and/or the avoidance of sexual intimacy.

Exclusion Criteria:

1. Urinary system infection: Abnormal result of routine urine and prostatic fluid routine examination;
2. Abnormal sex hormone: Abnormal result of sex hormone examination;
3. Systemic disease: hypertension, diabetes mellitus, alcohol dependence syndrome, coronary heart disease, and Mental disorder;
4. Organic disorder: Abnormal palpation of external genitals, testis, epididymis and spermatic cord;
5. Drug influence: use of any drug for PE, e.g. SSRI , PDE-5, tramadol, etc;
6. Known drug allergy to amide-type local anaesthetics or dapoxetine;
7. Currently participating, or in the past 30 days quit a another clinical research independent with this research;
8. Drugs, alcohol or substance abuse in last 6 months;
9. moderate or more severe erectile Dysfunction.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult males with sympton of premature ejaculation, excepting for other diseases.
Sampling Method: Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Intra-vaginal Ejaculation Latency Time（IELT） | After enrollment,after 4 weeks' treatment,after 8 weeks' treatment,after 12 weeks' treatment
  Most commonly used in research on premature ejaculation.
Change of score of Premature ejaculation diagnostic tool（PEDT） | After enrollment,after 12 weeks' treatment
  A questionnaire to evaluate and diagnose premature ejaculation
Change of grade Premature ejaculation profile（PEP） | After enrollment,after 4 weeks' treatment,after 8 weeks' treatment,after 12 weeks' treatment
  A questionnaire consists of 4 questions to evaluate the 4 aspects of the symptom of premature ejaculation
The change of results of Nerve electrophysiological examination | After enrollment,after 12 weeks' treatment
  To measure the penile sensory excitability and penile skin sympathetic excitability.
Clinical Global Impression of Change | After 12 weeks' treatment
  A single question to measure the change after treatment
Change of Chinese Index of Premature Ejaculation of five items(CIPE-5) | After enrollment,after 12 weeks' treatment
  A questionnaire to evaluate and diagnose premature ejaculation designed for Chinese people

CONTACTS AND LOCATIONS:
Overall Officials: Yutian Dai, Doctor, Study Chair — Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School
Locations (6):
- China (6):
  - Jingling Hospital, Nanjing, Jiangsu
  - Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu

REFERENCES:
- [Background] Waldinger MD. Recent advances in the classification, neurobiology and treatment of premature ejaculation. Adv Psychosom Med. 2008;29:50-69. doi: 10.1159/000126624. PMID 18391557
- [Background] Waldinger MD. The neurobiological approach to premature ejaculation. J Urol. 2002 Dec;168(6):2359-67. doi: 10.1016/S0022-5347(05)64146-8. PMID 12441918
- [Background] Althof SE, McMahon CG, Waldinger MD, Serefoglu EC, Shindel AW, Adaikan PG, Becher E, Dean J, Giuliano F, Hellstrom WJ, Giraldi A, Glina S, Incrocci L, Jannini E, McCabe M, Parish S, Rowland D, Segraves RT, Sharlip I, Torres LO. An Update of the International Society of Sexual Medicine's Guidelines for the Diagnosis and Treatment of Premature Ejaculation (PE). Sex Med. 2014 Jun;2(2):60-90. doi: 10.1002/sm2.28. PMID 25356302
- [Result] Serefoglu EC, McMahon CG, Waldinger MD, Althof SE, Shindel A, Adaikan G, Becher EF, Dean J, Giuliano F, Hellstrom WJ, Giraldi A, Glina S, Incrocci L, Jannini E, McCabe M, Parish S, Rowland D, Segraves RT, Sharlip I, Torres LO. An evidence-based unified definition of lifelong and acquired premature ejaculation: report of the second international society for sexual medicine ad hoc committee for the definition of premature ejaculation. Sex Med. 2014 Jun;2(2):41-59. doi: 10.1002/sm2.27. PMID 25356301
- [Result] McMahon CG, Althof SE, Waldinger MD, Porst H, Dean J, Sharlip ID, Adaikan PG, Becher E, Broderick GA, Buvat J, Dabees K, Giraldi A, Giuliano F, Hellstrom WJ, Incrocci L, Laan E, Meuleman E, Perelman MA, Rosen RC, Rowland DL, Segraves R. An evidence-based definition of lifelong premature ejaculation: report of the International Society for Sexual Medicine (ISSM) ad hoc committee for the definition of premature ejaculation. J Sex Med. 2008 Jul;5(7):1590-606. doi: 10.1111/j.1743-6109.2008.00901.x. PMID 18466262
- [Result] Dinsmore WW, Wyllie MG. PSD502 improves ejaculatory latency, control and sexual satisfaction when applied topically 5 min before intercourse in men with premature ejaculation: results of a phase III, multicentre, double-blind, placebo-controlled study. BJU Int. 2009 Apr;103(7):940-9. doi: 10.1111/j.1464-410X.2009.08456.x. Epub 2009 Feb 23. PMID 19245438
- [Result] McMahon CG. Efficacy of dapoxetine in the treatment of premature ejaculation. Clin Med Insights Reprod Health. 2011 Aug 2;5:25-39. doi: 10.4137/CMRH.S7337. eCollection 2011 Aug 2. PMID 24453509
- [Result] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176
- [Result] Xia JD, Zhou LH, Han YF, Chen Y, Wang R, Dai YT. A reassessment of penile sensory pathways and effects of prilocaine-lidocaine cream in primary premature ejaculation. Int J Impot Res. 2014 Sep-Oct;26(5):186-90. doi: 10.1038/ijir.2014.5. Epub 2014 Feb 27. PMID 24572995
- [Result] Xia JD, Han YF, Zhou LH, Xu ZP, Chen Y, Dai YT. Sympathetic skin response in patients with primary premature ejaculation. Int J Impot Res. 2014 Jan;26(1):31-4. doi: 10.1038/ijir.2013.23. Epub 2013 May 2. PMID 23636274
- [Result] Xia J, Chen T, Chen J, Han Y, Xu Z, Zhou L, Chen Y, Dai Y. The sympathetic skin response located in the penis as a predictor of the response to sertraline treatment in patients with primary premature ejaculation. J Sex Med. 2014 Nov;11(11):2801-8. doi: 10.1111/jsm.12654. Epub 2014 Aug 8. PMID 25130949